CLINICAL TRIAL: NCT05711355
Title: A Randomized Trial of the Effects of Platelet-Rich Plasma on Postoperative Complications After Meningomyelocele Sac Repair
Brief Title: the Effects of Platelet-Rich Plasma on Postoperative Complications After Meningomyelocele
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yuzuncu Yil University (Other)
Responsible Party: Principal Investigator, Özkan Arabaci, assosiation professor, Yuzuncu Yil University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: YuzuncuYıl1
Record Dates: First submitted 2022-12-09; First posted 2023-02-03 (Actual); Last update posted 2023-02-03 (Actual); Status verified 2023-01

CONDITIONS: Meningomyelocele/Spina Bifida
Keywords: Meningomyelocele; myelomeningocele; neural tube defect; spina bifida; platelet-rich plasma; cerebrospinal fluid
MeSH Terms: conditions — Meningomyelocele; Spinal Dysraphism; Neural Tube Defects

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Use of Platelet-Rich Plasma after meningomyelocele sac repair (Active Comparator): Paitents treated with platelet-rich plasma injection and treated with according to guidelines
  Interventions: Procedure: Use of Platelet-Rich Plasma after meningomyelocele sac repair; Procedure: meningomyelocele sac repair
- Control group of meningomyelocele sac repair (Active Comparator): Paitents treated according to guidelines
  Interventions: Procedure: meningomyelocele sac repair

INTERVENTIONS:
Procedure: Use of Platelet-Rich Plasma after meningomyelocele sac repair — Wound healing with the use of Platelet-Rich Plasma after surgical meningomyelocele pouch repair
  Arms: Use of Platelet-Rich Plasma after meningomyelocele sac repair
Procedure: meningomyelocele sac repair — meningomyelocele sac repair without Platelet-Rich Plasma

SUMMARY:
Introduction: Meningomyelocele is a common congenital neural tube defect. To reduce complications, early surgery and a multidisciplinary approach is needed. In this study, the investigators administered platelet-rich plasma (PRP) to newborns with meningomyelocele following corrective surgery to minimize cerebrospinal fluid (CSF) leakage and accelerate the healing of the immature pouch tissue. The investigators compared these with a control group that did not receive PRP.

Patients and Methods: Of the 40 newborns who were operated on with the diagnosis of meningomyelocele, 20 patients received PRP after surgical repair, and 20 were followed up without PRP. In the PRP group, 10 of the 20 patients underwent primary defect repair, the other 10 underwent flap repair. In the group that did not receive PRP, primary closure was performed in 14 patients and flap closure in six.

DETAILED DESCRIPTION:
Introduction Meningomyelocele (MMC), a form of spina bifida, is the most common congenital anomaly of the central nervous system. It occurs in the first four weeks of pregnancy when the neural tube of the embryo fails to close. Neural tube defects may result in hydrocephalus, hindbrain herniation, and exposure to toxins in the amniotic fluid, with potential morbidity and mortality (1). Both environmental and genetic factors contribute to the etiology of MMC. The risk of MMC is increasing in the events of maternal exposure to valproate, alcohol, carbamazepine, or isotretinoin; high fever; malnutrition, especially folate or B12 deficiency, diabetes mellitus, or obesity during pregnancy (2). About 1,427 babies are born with spina bifida each year in the United States (1 in 2,758 births). Lower socioeconomic status and older maternal age are associated with higher neural tube defect incidence. The recurrence rate in subsequent pregnancies is about 2% to 3% (3). More than 80% of babies born with MMC require a ventriculoperitoneal shunt for hydrocephalus decompression (4). In 39% of the patients, functional motor deficits are at the affected level or higher, and more than half of these have functional motor deficits two levels higher than the affected level (5). The purpose of early closure of MMC defects is to preserve neural tissue function and prevent sepsis.

Platelet-rich plasma (PRP) is an autologous concentration of human platelets obtained from venous blood through proper centrifugation. It contains several growth factors including platelet-derived growth factor (PDGF), vascular endothelial growth factor (VEGF), epidermal growth factor (EGF), platelet-derived factor 4 (PF-4), insulin-like growth factor (IGF-1), and transforming growth factor-beta (TGF-b) (6). There are approximately 150-400 10³/mm³ platelets in the blood and PRP contains between four and seven times this amount (7). When whole blood is collected from a patient for the generation of PRP, an anticoagulant is added. This usually contains citrate and disrupts the coagulation cascade by binding to calcium ions (8). PRP is used in orthopedic indications, wound healing, facial rejuvenation, hair restoration, and other conditions in which tissue renewal is central. The use of PRP for surgical and non-surgical wounds is advantageous, especially in patients with poor wound healing, poor blood supply, and slow cell turnover, and in cases where rapid healing is required.

In this study, we assessed whether the administration of PRP during the MMC pouch repair procedure can improve infant outcomes. This was measured by its ability to reduce CSF leakage, meningitis, local infection, skin necrosis, wound dehiscence, and hydrocephalus, and to accelerate the healing of the underdeveloped pouch tissue. These outcomes were compared with those of an MMC control group who did not receive PRP during surgery.

Materials and Methods This study included 40 infants with a diagnosis of MMC who were operated on at our neurosurgery clinic between February 2020 and May 2021. PRP was administered to 20 of the patients and 20 were followed up without PRP. All babies were born at term and fed with breast milk. All infants in the study were followed up in the neonatal intensive care unit. The mean birth weight was 2990 grams. In the PRP group, 10 of the 20 patients underwent primary defect repair and 10 underwent flap repair. In the non-PRP group, 14 patients underwent primary closure and six underwent flap closure. All operations were performed under general anesthesia. Blood was taken from each patient and the platelets were separated by centrifugation at 3200 rpm for five min in a 2 cc whole blood centrifuge device. The plasma was separated with the buffy coat layer. During MMC sac repair, a neural plate was formed and the dura was then made using opposing flaps from the fascia. After hemostasis was achieved, the defect was repaired and PRP was applied from the wound edge. The prepared PRP was applied to the dura and pouch repair and under the skin flap wound line.

Descriptive statistics were expressed as means, standard deviations, medians, ranges, frequencies, and ratios. The distribution of variables was measured with the Kolmogorov-Smirnov test. Independent sample t-tests and Mann-Whitney U tests were used for the analysis of quantitative independent data. Chi-square tests were used in the analysis of qualitative independent data, and the Fischer test was used when the chi-square test conditions were not met. Analyses were performed using SPSS 27.0 software.

ELIGIBILITY:
Inclusion Criteria:

* Newborn babies born with a meningomyelocele sac

Exclusion Criteria:

* Newborn babies without a meningomyelocele sac

Ages: 1 Day to 1 Month | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2022-01-15 (Actual); Primary Completion 2022-11-15 (Actual); Study Completion 2022-12-15 (Actual)

PRIMARY OUTCOMES:
Skin Dehicense Occurrence | up to first 14 days after the surgery
  Area of surgery has been examined daily for skin dehisence
Partial Skin Necrosis Occurrence | up to first 14 days after the surgery
  Area of surgery has been examined daily for skin necrosis
CSF Leak Occurrence | up to first 14 days after the surgery
  Area of surgery has been examined daily for CSF leakage
Local Infection Occurrence | up to first 14 days after the surgery
  Area of surgery has been examined daily for wound infection

SECONDARY OUTCOMES:
Hydrocephalus Occurrence | birth to 6 months
  Patients had examined as out-patients monthly for 6 months with head circumference documentation and with cranial MRIs

CONTACTS AND LOCATIONS:
Overall Officials: Mehmet Edip Akyol, Ass. Prof, Study Director — Van Yuzuncu Yıl Unıversty
Locations (1):
- Van Yuzuncu Yıl Unıversty, Van, Turkey (Türkiye)

REFERENCES:
- [Background] Moldenhauer JS, Adzick NS. Fetal surgery for myelomeningocele: After the Management of Myelomeningocele Study (MOMS). Semin Fetal Neonatal Med. 2017 Dec;22(6):360-366. doi: 10.1016/j.siny.2017.08.004. Epub 2017 Oct 12. PMID 29031539
- [Background] Sahni M, Alsaleem M, Ohri A. Meningomyelocele(Archived). 2023 Sep 4. In: StatPearls [Internet]. Treasure Island (FL): StatPearls Publishing; 2025 Jan-. Available from http://www.ncbi.nlm.nih.gov/books/NBK536959/ PMID 30725644
- [Background] Mai CT, Isenburg JL, Canfield MA, Meyer RE, Correa A, Alverson CJ, Lupo PJ, Riehle-Colarusso T, Cho SJ, Aggarwal D, Kirby RS; National Birth Defects Prevention Network. National population-based estimates for major birth defects, 2010-2014. Birth Defects Res. 2019 Nov 1;111(18):1420-1435. doi: 10.1002/bdr2.1589. Epub 2019 Oct 3. PMID 31580536
- [Background] Rintoul NE, Sutton LN, Hubbard AM, Cohen B, Melchionni J, Pasquariello PS, Adzick NS. A new look at myelomeningoceles: functional level, vertebral level, shunting, and the implications for fetal intervention. Pediatrics. 2002 Mar;109(3):409-13. doi: 10.1542/peds.109.3.409. PMID 11875133
- [Background] Cochrane DD, Wilson RD, Steinbok P, Farquharson DF, Irwin B, Irvine B, Chambers K. Prenatal spinal evaluation and functional outcome of patients born with myelomeningocele: information for improved prenatal counselling and outcome prediction. Fetal Diagn Ther. 1996 May-Jun;11(3):159-68. doi: 10.1159/000264297. PMID 8739582
- [Background] Araki J, Jona M, Eto H, Aoi N, Kato H, Suga H, Doi K, Yatomi Y, Yoshimura K. Optimized preparation method of platelet-concentrated plasma and noncoagulating platelet-derived factor concentrates: maximization of platelet concentration and removal of fibrinogen. Tissue Eng Part C Methods. 2012 Mar;18(3):176-85. doi: 10.1089/ten.TEC.2011.0308. Epub 2011 Nov 22. PMID 21951067
- [Background] Alves R, Grimalt R. A Review of Platelet-Rich Plasma: History, Biology, Mechanism of Action, and Classification. Skin Appendage Disord. 2018 Jan;4(1):18-24. doi: 10.1159/000477353. Epub 2017 Jul 6. PMID 29457008
- [Background] Marx RE. Platelet-rich plasma (PRP): what is PRP and what is not PRP? Implant Dent. 2001;10(4):225-8. doi: 10.1097/00008505-200110000-00002. No abstract available. PMID 11813662
- [Background] Tamburrini G, Frassanito P, Iakovaki K, Pignotti F, Rendeli C, Murolo D, Di Rocco C. Myelomeningocele: the management of the associated hydrocephalus. Childs Nerv Syst. 2013 Sep;29(9):1569-79. doi: 10.1007/s00381-013-2179-4. Epub 2013 Sep 7. PMID 24013327
- [Background] Shaer CM, Chescheir N, Schulkin J. Myelomeningocele: a review of the epidemiology, genetics, risk factors for conception, prenatal diagnosis, and prognosis for affected individuals. Obstet Gynecol Surv. 2007 Jul;62(7):471-9. doi: 10.1097/01.ogx.0000268628.82123.90. PMID 17572919
- [Background] Oncel MY, Ozdemir R, Kahilogullari G, Yurttutan S, Erdeve O, Dilmen U. The effect of surgery time on prognosis in newborns with meningomyelocele. J Korean Neurosurg Soc. 2012 Jun;51(6):359-62. doi: 10.3340/jkns.2012.51.6.359. Epub 2012 Jun 30. PMID 22949965
- [Background] McLone DG. Care of the neonate with a myelomeningocele. Neurosurg Clin N Am. 1998 Jan;9(1):111-20. PMID 9405769
- [Background] Messing-Junger M, Rohrig A. Primary and secondary management of the Chiari II malformation in children with myelomeningocele. Childs Nerv Syst. 2013 Sep;29(9):1553-62. doi: 10.1007/s00381-013-2134-4. Epub 2013 Sep 7. PMID 24013325
- [Background] Mummareddy N, Dewan MC, Mercier MR, Naftel RP, Wellons JC 3rd, Bonfield CM. Scoliosis in myelomeningocele: epidemiology, management, and functional outcome. J Neurosurg Pediatr. 2017 Jul;20(1):99-108. doi: 10.3171/2017.2.PEDS16641. Epub 2017 Apr 28. PMID 28452655
- [Background] Wu PI, Diaz R, Borg-Stein J. Platelet-Rich Plasma. Phys Med Rehabil Clin N Am. 2016 Nov;27(4):825-853. doi: 10.1016/j.pmr.2016.06.002. PMID 27788903
- [Background] Nguyen RT, Borg-Stein J, McInnis K. Applications of platelet-rich plasma in musculoskeletal and sports medicine: an evidence-based approach. PM R. 2011 Mar;3(3):226-50. doi: 10.1016/j.pmrj.2010.11.007. PMID 21402369
- [Background] Rehman L, Shiekh M, Afzal A, Rizvi R. Risk factors, presentation and outcome of meningomyelocele repair. Pak J Med Sci. 2020 Mar-Apr;36(3):422-425. doi: 10.12669/pjms.36.3.1237. PMID 32292446
- [Background] Demir N, Peker E, Gulsen I, Agengin K, Tuncer O. Factors affecting infection development after meningomyelocele repair in newborns and the efficacy of antibiotic prophylaxis. Childs Nerv Syst. 2015 Aug;31(8):1355-9. doi: 10.1007/s00381-015-2701-y. Epub 2015 Apr 14. PMID 25870027
- [Background] Lien SC, Maher CO, Garton HJ, Kasten SJ, Muraszko KM, Buchman SR. Local and regional flap closure in myelomeningocele repair: a 15-year review. Childs Nerv Syst. 2010 Aug;26(8):1091-5. doi: 10.1007/s00381-010-1099-9. Epub 2010 Mar 2. PMID 20195618